CLINICAL TRIAL: NCT00651001
Title: Prevalence of Cardiovascular Risk Factors in Minorca - Spain
Brief Title: Metabolic Syndrome and Leptin Level Associated With Fructose Consumption in Spain
Status: Completed | Type: Observational
Sponsor: Hospital Mateo Orfila (Other)
Responsible Party: Perez-Pozo, Santos E. Lopez-Lillo, Julian. Johnson, Richard, Hospital Mateo Orfila, University of Florida
Other Study IDs: IbSalut-M-002
Record Dates: First submitted 2008-03-28; First posted 2008-04-02 (Estimated); Last update posted 2009-08-06 (Estimated); Status verified 2009-08

CONDITIONS: Healthy
Keywords: fructose; leptin; metabolic syndrome; blood pressure; inflammation; Relationship of fructose intake to leptin levels; Relationship of fructose to metabolic syndrome; Relationship of fructose to inflammation parameters; Relationship of fructose to blood pressure
MeSH Terms: conditions — Metabolic Syndrome; Inflammation

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum and urine collections.
Oversight: Data Monitoring Committee: No

SUMMARY:
A Food Frequency Questionnaire (FFQ), will be provided to 800 adults to assess overall fructose intake and this will be related to a number of features related to the metabolic syndrome, including serum leptin, characteristic features of metabolic syndrome (body mass index, waist circumference, plasma lipids, blood pressure, HOMA index,fasting glucose and fasting insulin levels) and other as: CRP, fibrinogen, homocysteine and uric acid.

ELIGIBILITY:
Inclusion Criteria:

* Adults, 18-70 years of age

Exclusion Criteria:

* Diabetes
* Kidney Failure
* Heart Failure
* Cancer

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 800 Adults, age 18 to 70
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2008-06; Primary Completion 2009-01 (Actual); Study Completion 2009-06

PRIMARY OUTCOMES:
Serum leptin levels as it relates to fructose intake | Epidemiological association

SECONDARY OUTCOMES:
Relationship of metabolic syndrome features with fructose intake. This includes measuring all 5 components of metabolic syndrome, assessing insulin resistance by HOMA, and measuring some markers of inflammation (CRP, fibrinogen, homocysteine) | Epidemiological

CONTACTS AND LOCATIONS:
Locations (1):
- Renal Unit of Mateo Orfila Hospital, Balearic Islands - Spain, Menorca, Balearic Islands, Spain